CLINICAL TRIAL: NCT05998850
Title: Community Health Worker Navigation of Community Resources for Dialysis Patients: A Pilot Intervention
Brief Title: Dialysis CHW Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Tessa Novick, Assistant Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00004663
Record Dates: First submitted 2023-07-19; First posted 2023-08-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Diseases; RENAL INSUFFICIENCY, CHRONIC
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Health Resources

STUDY DESIGN:
Intervention Model Description: IMPaCT (Individualized Management for Patient-Centered Targets)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CHW Dialysis Implementation (Experimental): A single-arm 6-month pilot study testing the feasibility of tailored implementation, by using IMPaCT model with a Community Health Worker to help low-income dialysis patient to navigate the health system and community resources to eliminate or minimize health-related social needs among dialysis patients so that they adhere to the treatment, improve their health and may be candidates for transplantation.
  Interventions: Behavioral: Community Health Worker Support with Resources

INTERVENTIONS:
Behavioral: Community Health Worker Support with Resources — 6-months of hands-on tailored support spanning the domains of social support, advocacy and navigation to achieve their action plans.

SUMMARY:
To determine the acceptability and feasibility of a community health worker intervention that assists dialysis patients with low socioeconomic status navigate community resources to address health-related social needs. Findings will be used for a future randomized trial that determines the efficacy of the CHW intervention on mental health, quality of life, addressing social needs, and clinical outcomes. This study is intended to be generalizable in all dialysis centers.

DETAILED DESCRIPTION:
The research team will conduct a single-arm 6-month pilot study testing the feasibility of implementing a tailored, health-related social needs intervention among dialysis patients. The research teamwill recruit 30 dialysis (all modalities) patients aged≥18 years with low socioeconomic status to participate in a CHW intervention. The CHW intervention will be modeled after IMPaCT (Individualized Management for Patient-Centered Targets), a 6-month CHW intervention that addresses "upstream" socioeconomic and behavioral barriers to treatment for individuals with chronic diseases, which has been adapted to numerous populations and shown to improve care and reduce hospitalizations. The CHW will identify health-related social needs and help participants navigate community resources to meet needs. All participants will receive the intervention. All participants will also participate in a CHW-led support group, that will occur monthly. The research team will compare outcomes during the 6-months before and during the intervention period. This pilot study aims to (1) assess the feasibility of recruiting dialysis patients experiencing health-related social needs to an intervention trial, and (2) assess the feasibility of implementing the intervention within this population, in a fashion deemed acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Have kidney failure and be receiving dialysis

Exclusion Criteria:

* Live in a nursing facility or institution
* Physically or mentally unable or unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participant recruited and ended intervention | 1-year
  To measure Study Feasibility the research team will be assessing the number of participants enrolled and recruitment at the beginning of the intervention and the number of participants that engage by ending the intervention. These measurements will provide information on the feasibility of the intervention among low-income people receiving dialysis treatment.
Number of participants accepting the CWH intervention as helpful | 1-year
  Assess acceptability at follow-up with a focus group. All participants will complete a focus group that discusses: (1) whether the CHW's guidance/assistance was helpful in meeting needs; (2) the utility of having the CHW work with them outside of the dialysis unit; (3) the perceived knowledge of the CHW; (4) the perceived willingness and ability of community partners to participate in the intervention; (5) general satisfaction; and (6) input on the intervention design. This qualitative analysis on the acceptability of the intervention among the participants will provide us with data on which components of the intervention are feasible to improve the quality of life and health in the target population, and what type of components we should improve and/or change to increase the effectiveness of the intervention. acceptability.

SECONDARY OUTCOMES:
Number of participants changing levels of depression in pre-post test | 1-Year
  This study will not be powered to detect differences in outcomes. However, in order to estimate the needed sample size for a future trial, the research team will collect information on the following outcomes pre-post changes in symptoms of depression by using the Beck depression inventory. The research team is expecting in the future that the levels of depression will get lower or none after the intervention.
Number of participants changing levels of anxiety in pre-post | 1-Year
  This study will not be powered to detect differences in outcomes. However, in order to estimate the needed sample size for a future trial, the research team will collect information on the following outcomes pre-post changes in symptoms of anxiety by using GAD-7 Anxiety inventory. The research team is expecting in the future that the levels of anxiety will get lower or none after the intervention.
Number of participants changing levels of quality of life in pre-post | 1-Year
  This study will not be powered to detect differences in outcomes. However, in order to estimate the needed sample size for a future trial, the research team will collect information on the following outcomes pre-post changes in the quality of life. The research team is expecting in the future that the levels of better quality of life will get higher after the intervention.
Number of connection with community resources per participants in pre-post | 1-Year
  The research team is expecting a greater amount of connection made with a community resource after the intervention.
Number of dialysis session missed, ended early and amount of participants in transplanting listing. | 1-Year
  The research team is expecting less number of missed dialysis sessions, an increase in the number of times the participant ended a dialysis session early, and an increase of participants in transplant listing.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa K Novick, MSW, MD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will develop manuscripts and do presentations to release information and results.
Supporting Information: Study Protocol
Time Frame: The data will become available in 2025 and will be available for two years.